CLINICAL TRIAL: NCT03865329
Title: Increasing Adherence to Pulmonary Rehabilitation After COPD Related Hospitalizations
Brief Title: Increasing Adherence to Pulmonary Rehabilitation After COPD Related Hospitalizations (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-002453 (Pilot Study/R61); R61HL142933 (NIH)
Record Dates: First submitted 2019-01-21; First posted 2019-03-06 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention- Home Pulmonary Rehabilitation (Experimental): Participants will be offered a Home-based pulmonary rehabilitation program with health coaching.
  Interventions: Behavioral: Intervention- Home-based Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Intervention- Home-based Pulmonary Rehabilitation — Home-based Pulmonary Rehabilitation (PR) with health coaching using a remote system that will allow patients to complete PR at home. The program involves upper and lower extremity exercises, self-report of symptoms (fatigue, breathlessness, physical activity and overall well-being).

SUMMARY:
This pilot study will look at investigating barriers, facilitators, adherence and effectiveness of an interactive home-based pulmonary rehabilitation program and health coaching for patients who have recently been hospitalized for a COPD related cause.

DETAILED DESCRIPTION:
Despite proven benefits, the proportion of people with COPD who receive Pulmonary Rehabilitation (PR) is very small. The current model of a center-based PR program fails to address the needs of many patients with COPD. The most common patient barrier to attendance is travel to center-based programs, particularly for frail patients with more severe COPD who need transportation assistance. Home-based, unsupervised PR has been proposed as an alternative model to hospital-based programs and has been found to be safe and effective.

In this pilot study researchers will investigate barriers, facilitators and adherence to a home-based pulmonary rehabilitation program after hospitalization. The results of this pilot study will inform the second part of this study as a randomized control study under a different grant (Study 2/R33). Both quantitative and qualitative methods will be used for the evaluation.

10 patients will be enrolled in this pilot study and allocated to a home-based PR in order to polish the intervention before the randomized portion of the study. This pilot is supported by a grant mechanism (R61) explicitly oriented to adjust the intervention and identify barriers for the next randomized portion of this study (Study 2) supported by a separate grant mechanism (R33).

ELIGIBILITY:
Inclusion Criteria

* COPD related hospitalization and eligible for PR
* Age 40+
* Confidence (score > 5 in a self-efficacy question (1-10 scale): how confident you feel to use this system on a daily basis)

Exclusion Criteria

* Inability to walk (orthopedic-neurologic problems or confined to bed)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Adherence to One Balance Practice Routine
Description: Percentage of participants to adhere to one balance practice routine per day for 6 out of the 7 days for 12 weeks prescribed via the interactive home-based pulmonary rehabilitation program
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
percentage of participants | 49

2. Primary Outcome: Adherence to Two Balance Practice Routine
Description: Percentage of participants to adhere to two balance practices routine per day for 6 out of the 7 days for 12 weeks prescribed via the interactive home-based pulmonary rehabilitation program
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
percentage of participants | 42

3. Primary Outcome: Adherence to Daily Flexible Practice Routine
Description: Percentage of participants to adhere to the daily flexible practice routine for 6 out of the 7 days for 12 weeks prescribed via the interactive home-based pulmonary rehabilitation program
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
percentage of participants | 54

4. Primary Outcome: Completion of the Daily Self-assessment
Description: Percentage of participants to complete the daily self-assessment for 6 out of the 7 days for 12 weeks via the interactive home-based pulmonary rehabilitation program
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
percentage of participants | 61

5. Secondary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Physical Symptoms Summary
Description: The CRQ is a 20-question inventory assessing the areas of health related quality of life in dyspnea (shortness of breath), fatigue, emotion, and feelings of mastery of chronic respiratory disease. The Physical Summary score includes dyspnea (symptom #1 in COPD) and fatigue (symptom #2 in COPD) domains. The questions in each domain are added together and then divided by the number of questions. The possible range is 1-7, where 1 is the worst and 7 the best.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
score on a scale | 0.5 (1.6)
Statistical Analysis 1: Comparison: Intervention- Home Pulmonary Rehabilitation; Test type: Superiority; p = 0.13, t-test, 2 sided

6. Secondary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Emotional Symptoms Summary
Description: The CRQ Emotion Summary score includes the emotion (independent factor for admissions and poor quality of life) and mastery (self-management) domains of the CRQ. The scores for each domain are calculated by simply added together the answers and then dividing by the number of questions, the range is 1-7 where 1 is the worst and 7 the best.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
score on a scale | 0.6 (1.7)
Statistical Analysis 1: Comparison: Intervention- Home Pulmonary Rehabilitation; Test type: Superiority; p = 0.01, t-test, 2 sided

7. Secondary Outcome: Daily Physical Activity
Description: Average number of steps per day recorded by ActiGraph activity monitor worn on the wrist for seven days at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
steps | 4086.3 (2552.2)

8. Secondary Outcome: Change in the Self-Management Ability Scale (SMAS) Total Score
Description: Measured using the total score from the self-reported SMAS 30 item questionnaire that measures ability and function. A higher score indicates more ability and function in everyday life. The SMAS30 has six areas, each with 5 questions. The minimum score is one and the max is 5. The mean is calculated for each section. A higher score indicates better self management.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
score on a scale | 3.8 (13)
Statistical Analysis 1: Comparison: Intervention- Home Pulmonary Rehabilitation; Test type: Superiority; p = 0.10, t-test, 2 sided

9. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-2)
Description: Measured using the self-reported PHQ-2 consisting of a 2 item questionnaire inquiring about the frequency of depressed mood over the past 2 weeks on a scale of 0 to 3, 0=Not at all, 1=several days, 2=more than half the days, 3=nearly everyday. The minimum score is zero and the highest score is 6. A score greater than 3 may indicate depression.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation
Number analyzed (Participants) | 9
score on a scale | -0.6 (1.9)
Statistical Analysis 1: Comparison: Intervention- Home Pulmonary Rehabilitation; Test type: Superiority; p = 0.25, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 3 months on all participants.
Groups:
- Intervention- Home Pulmonary Rehabilitation: Home-based Pulmonary Rehabilitation (PR) with health coaching using a remote system that will allow patients to complete PR at home. The program involves upper and lower extremity exercises, self-report of symptoms (fatigue, breathlessness, physical activity and overall well-being).
  Intervention- Home-based Pulmonary Rehabilitation: Participants enrolled in the intervention arm will be offered a Home-based pulmonary rehabilitation program with health coaching.
Arm/Group | Intervention- Home Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03865329/Prot_SAP_000.pdf